CLINICAL TRIAL: NCT06436495
Title: Validation of Methodologies: Correlating Adherent Scalp Flaking Score (ASFS) With Phototrichogram for Comprehensive Evaluation of Scalp Dandruff in Adults
Brief Title: Methodology Validation: Correlating Adherent Scalp Flaking Score (ASFS) With Phototrichogram for Scalp Dandruff Evaluation in Adult Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Responsible Party: Principal Investigator, Maheshvari Patel, Principal Investigator - Director (Operations), NovoBliss Research Pvt Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NB240024-NB-V
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Dandruff
MeSH Terms: conditions — Dandruff

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Cohort (Experimental): The complete study group will be given hair-wash intervention post baseline evaluations.
  Interventions: Other: Hair Wash Shampoo

INTERVENTIONS:
Other: Hair Wash Shampoo — A standard marketed hair wash shampoo is to be used for the hair wash intervention post baseline evaluations of the scalp.
  Other Names: Dove Hair Wash Shampoo

SUMMARY:
This study aims to validate methods for assessing scalp hair dandruff by comparing three evaluation techniques: the Adherent Scalp Flaking Score (ASFS), Phototrichogram, and 60-second hair combing.

These assessments will be conducted before and after hair wash interventions on adult human subjects to evaluate adherent and non-adherent scalp flakes. By comparing the results of these evaluations, the study aims to determine the consistency and reliability of each method in assessing the presence and severity of dandruff. Establishing correlation between these assessment techniques is essential for validating their usefulness in evaluating the effectiveness of hair care products and treatments in reducing scalp dandruff. This research aims to improve the accuracy and reliability of dandruff evaluation methods, benefiting both dermatological research and clinical practice in managing this prevalent condition.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years (both inclusive).
* Good general health as determined from recent medical history.
* No previous history of adverse skin conditions, and not under any medication likely to interfere with the results.

Exclusion Criteria:

* Non-willing subjects and subjects with a history of allergies or specific allergic reactions upon using dermatological/cosmetic products will not be included.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Adherent Scalp Flaking Score | On Day 1 - pre hair wash, and post hair wash and drying at T30 minutes.
  The score will be assessed by Dermatological Evaluation using the scoring scale where 0 indicates no flakes and 10 indicates heavy flakes
Scalp Condition using Phototrichogram | On Day 1 - pre hair wash, and post hair wash and drying at T30 minutes.
  The phototrichogram will be captured using CASLite Nova

SECONDARY OUTCOMES:
Non-adherent scalp flakes evaluation | On Day 1 - pre hair wash, and post hair wash and drying at T30 minutes.
  The assessment will be done via 60-second hair combing methods by dermatological assessment using 4 point scoring scale where 0=indicates none and 3 indicates heavy flakes

CONTACTS AND LOCATIONS:
Locations (1):
- NovoBliss Research Pvt Ltd, Gandhinagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: No